CLINICAL TRIAL: NCT04426058
Title: Complete Motor Sparing Protocol Versus Fascia Iliaca Suprainguinal Technique for Total Hip Arthroplasty, a Prospective Randomized Clinical Trial.
Brief Title: CMP vs Fascia Iliaca Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Scott Byram MD, MD, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213048
Record Dates: First submitted 2020-05-13; First posted 2020-06-11 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Pain, Postoperative; Hip Arthroplasty
Keywords: Nerve Block; Fascia Iliaca Nerve Block; Complete Motor Sparing Protocol; Hip Arthroplasty; Pain control
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Cytidine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMP (Experimental): Cluneal nerve Block 0.25% bupivacaine 20ml Pericapsular Nerve group block 0.25% Bupivacaine 20ml Lateral femoral cutaneous Block 0.25% bupivacaine 10ml
  Interventions: Drug: CMP
- Fascia iliaca (Active Comparator): Fascia iliaca block suprainguinal technique 0.25% bupivacaine 50ml
  Interventions: Drug: Fascia Illica

INTERVENTIONS:
Drug: CMP — Cluneal nerve Block 0.25% bupivacaine 20ml Pericapsular Nerve group block 0.25% Bupivacaine 20ml Lateral femoral cutaneous Block 0.25% bupivacaine 10ml
  Arms: CMP
Drug: Fascia Illica — Fascia iliaca block suprainguinal technique 0.25% bupivacaine 50ml
  Arms: Fascia iliaca

SUMMARY:
Complete motorsparing protocol (CMP) has been developed to try to minimize the motor nerve block that is created when using Facia iliaca nerve block. The blocks performed in the (CMP) are the cluneal nerve block, Pericapsular nerve group block and lateral femoral cutaneous block. On the clinical trial, the investigators will randomize the participants that meet criteria to CMP or Fascia iliaca Block and compare the amount of opioid needed post op during 24 hours and their pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients undergoing total hip arthroplasty posterior approach.
* Patients willing to participate and sign informed consent

Exclusion Criteria:

* Severe COPD/other contraindication to general anesthesia that spinal would be more suitable.
* Patient with a weight of less than 41 kg
* Dementia, not alert or Oriented to person, place, or time
* Chronic pain patient with daily opioid use at home.
* Patient with allergy to local anesthetics
* Patient refusal
* Total hip arthroplasty revision
* Concomitant pain in different area from operative site.
* Pregnancy
* Patient with active infection on the injection sites for the blocks
* Patients unable or willing to understand or comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of opioid use | 24 hours
  Measurement of opioid use (mg) for pain control after surgery once patient in recovery area

SECONDARY OUTCOMES:
Measurement of the pain control | 24 hours
  Measurement of the pain control via numeric rating scale 0-10 where 0 is no pain and 10 is the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tyagi A, Salhotra R. Total hip arthroplasty and peripheral nerve blocks: Limited but salient role? J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):379-380. doi: 10.4103/joacp.JOACP_114_18. No abstract available. PMID 30386023
- [Background] Adhikary SD, Short AJ, El-Boghdadly K, Abdelmalak MJ, Chin KJ. Transmuscular quadratus lumborum versus lumbar plexus block for total hip arthroplasty: A retrospective propensity score matched cohort study. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):372-378. doi: 10.4103/joacp.JOACP_335_17. PMID 30386022
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Hannon CP, Keating TC, Lange JK, Ricciardi BF, Waddell BS, Della Valle CJ. Anesthesia and Analgesia Practices in Total Joint Arthroplasty: A Survey of the American Association of Hip and Knee Surgeons Membership. J Arthroplasty. 2019 Dec;34(12):2872-2877.e2. doi: 10.1016/j.arth.2019.06.055. Epub 2019 Jul 8. PMID 31371038
- [Background] Kumar K, Pandey RK, Bhalla AP, Kashyap L, Garg R, Darlong V, Malhotra R, Yadav CS. Comparison of conventional infrainguinal versus modified proximal suprainguinal approach of Fascia Iliaca Compartment Block for postoperative analgesia in Total Hip Arthroplasty. A prospective randomized study. Acta Anaesthesiol Belg. 2015;66(3):95-100. PMID 26767235
- See also: Randomized trial of ultrasound-guided superior cluneal nerve block — https://rapm.bmj.com/content/early/2019/05/16/rapm-2018-100174?versioned=true

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT04426058/Prot_000.pdf
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT04426058/ICF_001.pdf